CLINICAL TRIAL: NCT01752556
Title: Non-inferiority Randomized Control Trial About Efficacy and Cost-effectiveness of Home Respiratory Polygraphy Management in Sleep Apneas/Hypopneas Syndrome
Brief Title: Cost-effectiveness of Home Respiratory Polygraphy
Acronym: HRP-M
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Principal Investigator, Juan F. Masa, MD, Sociedad Española de Neumología y Cirugía Torácica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI12/01240
Record Dates: First submitted 2012-05-17; First posted 2012-12-19 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2016-12

CONDITIONS: Sleep Apnea Syndrome
Keywords: Sleep apnea, Portable monitor,autoCPAP
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hospital diagnosis (Active Comparator): diagnosis of Sleep Apnea and therapeutic decision will perform according to polysomnography
  Interventions: Procedure: diagnosis and therapeutic decision
- Home diagnosis (Experimental): diagnosis of Sleep Apnea and therapeutic decision will be perform according to home respiratory polygraphy
  Interventions: Procedure: diagnosis and therapeutic decision

INTERVENTIONS:
Procedure: diagnosis and therapeutic decision — A conventional polysomnography will be done to perform the diagnosis and therapeutic decision(CPAP or not). Treated and untreated will be followed 6 moths
  Arms: Hospital diagnosis
Procedure: diagnosis and therapeutic decision — A home respiratory polygraphy will be done to perform the diagnosis and therapeutic decision(CPAP or not). Treated and untreated will be followed 6 months
  Arms: Home diagnosis

SUMMARY:
Primary objectives:

The efficacy of the therapeutic decision taken by respiratory polygraphy (RP) against polysomnography (PSG) using the Epworth scale;

Secondary Objective:

1. the cost-effectiveness of diagnosis and therapeutic decision valued using the Epworth Scale and EuroQol 5D.
2. effectiveness of the therapeutic decision by means of: 1) quality of life tests, 2) adherence and compliance to treatment, 3) blood pressure MAP, 4) biochemistry determinations. Design: prospective, randomized, controlled, open, parallel of non-inferiority. 440 patients will be randomized to diagnose and follow treatment based on the RP or the PSG. The follow-up will last 6 months with 4 assessments. Statistical analysis: We will compare the change in the Epworth scale between both arms of treatment through analysis of covariance. The premise of non-inferiority is -2 at the lower limit of 95% IC. Secondary variables will be analyzed using differences in independent means (or non-parametric equivalent) or Chi2 for dichotomous variables. Cost-effectiveness: costs generated by one and another method will be evaluated against the effectiveness of the primary variable using Bayesian techniques

DETAILED DESCRIPTION:
Design: Prospective, randomized, controlled, open, parallel noninferiority. 440 patients will be randomized to diagnose and follow treatment based on the PR or PSG generating four groups: two treated and two untreated with CPAP. The latter did not undergo self-certification home. The monitoring will be 6 months and 4 assessments. Statistical analysis: compare the change of the scale Epworth before and after the intervention between both treatment arms using analysis of covariance. The premise is non-inferiority of -1.6 at the lower limit of 95%. Secondary variables were analyzed by independent means differences (or nonparametric equivalent) or Chi2 for dichotomous variables. Cost-effectiveness: the costs generated by the two methods will be measured against the effectiveness of the primary endpoint using Bayesian techniques

ELIGIBILITY:
Inclusion criteria:

1. Snoring or sleep apneas observed by partner
2. Symptoms that may be secondary to the apneas/hypopneas - concretely, an ESS ≥10
3. Age between 18 and 70
4. Absence of clinical suspicion of any other sleep pathology which could cause daytime sleepiness

Exclusion criteria:

1. Psycho-physical inability to complete questionnaires
2. documented structural or coronary cardiopathy not controlled by medical treatment
3. Cheyennes-Stokes Syndrome
4. Patient has undergone an uvulopalatopharyngoplasty
5. Unable to provide informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2012-05; Primary Completion 2015-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Determine the efficacy of diagnosis and therapeutic decision-making evaluated using Epworth sleepiness scale as primary variable in patients managed by home RP and by PSG after six months of follow-up. | Six months

SECONDARY OUTCOMES:
the cost-effectiveness of diagnosis and therapeutic decision valued using the Epworth Scale and EuroQol 5D. | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Juan F. Masa, MD, Principal Investigator — Hospital San Pedro de Alcántara. Cáceres. Spain
Locations (1):
- Juan F. Masa, Cáceres, Cáceres, Spain

REFERENCES:
- [Derived] Corral J, Sanchez-Quiroga MA, Carmona-Bernal C, Sanchez-Armengol A, de la Torre AS, Duran-Cantolla J, Egea CJ, Salord N, Monasterio C, Teran J, Alonso-Alvarez ML, Munoz-Mendez J, Arias EM, Cabello M, Montserrat JM, De la Pena M, Serrano JC, Barbe F, Masa JF; Spanish Sleep Network. Conventional Polysomnography Is Not Necessary for the Management of Most Patients with Suspected Obstructive Sleep Apnea. Noninferiority, Randomized Controlled Trial. Am J Respir Crit Care Med. 2017 Nov 1;196(9):1181-1190. doi: 10.1164/rccm.201612-2497OC. PMID 28636405